CLINICAL TRIAL: NCT04258839
Title: A Phase 3, Multicenter, Open Label Trial to Evaluate the Long-term Safety and Tolerability of Brexpiprazole in Treatment of Children and Adolescents With Irritability Associated With Autism Spectrum Disorder
Brief Title: Brexpiprazole in Treatment of Children and Adolescents With Irritability Associated With Autism Spectrum Disorder for Subjects That Have Completed Participation in 331-201-00148
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Collaborators: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 331-201-00191; 2018-004899-35 (EudraCT Number)
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Results first posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Irritability Associated With Autism Spectrum Disorder
Keywords: Autism; Autism Spectrum Disorder; ASD; Irritability
MeSH Terms: conditions — Autistic Disorder; Autism Spectrum Disorder | interventions — brexpiprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Brexpiprazole (Experimental): Participants received brexpiprazole based on the body weight for 26 weeks in this study.
  Participants with body weight < 50 kilograms (kg), received brexpiprazole tablets orally, once daily (QD) at dose of 0.25 mg on Days 1 to 3 followed by 0.5 mg on Days 4 to 7 and 1 mg on Days 8 to 14. Based on the investigator's judgment, the dose was increased to 1 or 1.5 mg starting from Day 15 until week 26.
  Participants with body weight ≥ 50 kg received brexpiprazole tablet orally, QD at dose of 0.5 mg on Days 1 to 3, followed by 1.5 mg on Days 4 to 7, and 2 mg on Days 8 to 14. Based on the investigator's judgment the dose was increased to 1.5, 2, or 3 mg starting from Day 15 until week 26.
  Interventions: Drug: Brexpiprazole

INTERVENTIONS:
Drug: Brexpiprazole — Oral tablet; taken once daily
  Other Names: OPC-34712; LuAF41156

SUMMARY:
The purpose of this study is to evaluate the long-term safety and tolerability of brexpiprazole in children and adolescent participants, aged 5 to 17, with irritability associated with autism spectrum disorder.

ELIGIBILITY:
Inclusion Criteria:

* 5 to 17 year of age or turned 18 while enrolled in the 331-201-00148 study
* Autism Spectrum Disorder
* Completion of 331-201-00148 trial
* Investigator assessment

Exclusion Criteria:

* Did not complete treatment period or incurred significant protocol deviations during 331-201-00148 study
* Sexually active males or female of childbearing potential who do not agree to practice 2 different methods of birth control or remain abstinent during the trial and for 30 days after the last dose
* Female with positive pregnancy test

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 95 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-03-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (28):
- United States (28):
  - Dothan Behavioral Medicine Clinic, Dothan, Alabama
  - Southwest Autism Research and Resource Center, Phoenix, Arizona
  - University of California San Francisco, Nancy Friend Pritzker Psychiatry, San Francisco, California
  - APG Research, Orlando, Florida
  - Autism Assessment, Research, Treatment and Services (AARTS) center, Chicago, Illinois
  - Research site, Lake Charles, Louisiana
  - The Lurie Center for Autism, Lexington, Massachusetts
  - Research site, Bloomfield Hills, Michigan
  - Thompson Center for Autism and Neurodevelopment, Columbia, Missouri
  - Research site, Saint Charles, Missouri
  - Alivation, Lincoln, Nebraska
  - Center for Psychiatry and Behavioral Medicine Inc., Las Vegas, Nevada
  - Rutger's-New Jersey Medical Scholl Clinical Research Unit, Newark, New Jersey
  - For additional information regarding sites, Princeton, New Jersey
  - Bioscience Research, Mount Kisco, New York
  - Research site, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - Research Site, Avon Lake, Ohio
  - The Holloway Group, Inc, Oklahoma City, Oklahoma
  - Access Clinical Trials, Nashville, Tennessee
  - Research site, Austin, Texas
  - Cedar Health Research, Dallas, Texas
  - Research site, San Antonio, Texas
  - UT Health San Antonio Long School of Medicine, Department of Psychiatry and Behavioral Sciences, San Antonio, Texas
  - Family Psychiatry of the Woodlands, The Woodlands, Texas
  - Woodstock Research Center, Woodstock, Vermont
  - Core Clinical Research, Everett, Washington

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com
URL: https://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with irritability associated with autism spectrum disorder (ASD) were enrolled in the study at sites in the United States from 23 January 2020 to 16 March 2023.
Pre-assignment Details: A total of 95 eligible participants who completed 8-week, double-blind treatment, in the parent study 331-201-00148 (NCT04174365) and, who in the investigator's judgment, could potentially benefit from receiving brexpiprazole were enrolled in this study. Data was summarized as per the treatment received in the parent study 331-201-00148 (NCT04174365).
Groups:
- Prior Brexpiprazole: Participants who received brexpiprazole in the parent study 331-201-00148 (NCT04174365) received brexpiprazole based on the body weight for 26 weeks in this study.
  Participants with body weight < 50 kilograms (kg), received brexpiprazole tablets orally, once daily (QD) at dose of 0.25 mg on Days 1 to 3 followed by 0.5 mg on Days 4 to 7 and 1 mg on Days 8 to 14. Based on the investigator's judgment, the dose was increased to 1 or 1.5 mg starting from Day 15 until week 26.
  Participants with body weight ≥ 50 kg received brexpiprazole tablet orally, QD at dose of 0.5 mg on Days 1 to 3, followed by 1.5 mg on Days 4 to 7, and 2 mg on Days 8 to 14. Based on the investigator's judgment the dose was increased to 1.5, 2, or 3 mg starting from Day 15 until week 26.
- Prior Placebo: Participants who received placebo matched to brexpiprazole in the parent study 331-201-00148 (NCT04174365) received brexpiprazole based on the body weight for 26 weeks in this study.
  Participants with body weight < 50 kg, received brexpiprazole tablets orally, QD at dose of 0.25 mg on Days 1 to 3 followed by 0.5 mg on Days 4 to 7 and 1 mg on Days 8 to 14. Based on the investigator's judgment, the dose was increased to 1 or 1.5 mg starting from Day 15 until week 26.
  Participants with body weight ≥ 50 kg received brexpiprazole tablet orally, QD at dose of 0.5 mg on Days 1 to 3, followed by 1.5 mg on Days 4 to 7, and to 2 mg on Days 8 to 14. Based on the investigator's judgment the dose was increased to 1.5, 2 or 3 mg starting from Day 15 until week 26.
Period: Overall Study
Arm/Group | Prior Brexpiprazole | Prior Placebo
Started | 49 | 46
Safety Sample (Safety Sample included all enrolled participants who received at least one dose of investigational medicinal product (IMP).) | 49 | 46
Efficacy Sample (Efficacy Sample included all participants in the Safety Sample who had a baseline assessment and at least one post-baseline assessment of the Aberrant Behavior Checklist - Irritability (ABC-I) subscale score.) | 48 | 46
Completed | 39 | 31
Not Completed | 10 | 15
Not completed — Adverse Event | 2 | 4
Not completed — Lack of Efficacy | 0 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Withdrawal by Caregiver | 5 | 6
Not completed — Reason not Specified | 0 | 1

BASELINE CHARACTERISTICS:
Population: Enrolled Sample included participants who completed the double-blind treatment period of the parent study 331-201-00148 (NCT04174365) and who gave consent/assent for participation into this open-label study and who also met all the eligibility criteria for this study.
Groups:
- Prior Brexpiprazole: Participants who received brexpiprazole in the parent study 331-201-00148 (NCT04174365) received brexpiprazole based on the body weight for 26 weeks in this study.
  Participants with body weight < 50 kg, received brexpiprazole tablets orally, QD at dose of 0.25 mg on Days 1 to 3 followed by 0.5 mg on Days 4 to 7 and 1 mg on Days 8 to 14. Based on the investigator's judgment, the dose was increased to 1 or 1.5 mg starting from Day 15 until week 26.
  Participants with body weight ≥ 50 kg received brexpiprazole tablet orally, QD at dose of 0.5 mg on Days 1 to 3, followed by 1.5 mg on Days 4 to 7, and 2 mg on Days 8 to 14. Based on the investigator's judgment the dose was increased to 1.5, 2, or 3 mg starting from Day 15 until week 26.
- Total: Total of all reporting groups
Arm/Group | Prior Brexpiprazole | Prior Placebo | Total
Number analyzed (Participants) | 49 | 46 | 95
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.0 (3.1) | 10.0 (3.1) | 10.0 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 8 | 12
  Male | 45 | 38 | 83
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 8 | 14
  Not Hispanic or Latino | 43 | 38 | 81
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 37 | 38 | 75
  Race: Black or African American | 8 | 2 | 10
  Race: Asian | 1 | 3 | 4
  Race: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Race: Other | 3 | 2 | 5
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 41.6 (17.9) | 44.2 (18.3) | 42.9 (18.1)
Simpson Angus Scale (SAS) Score [Mean (Standard Deviation); unit: score on a scale] — SAS was used to evaluate extrapyramidal symptoms (EPS). The SAS consists of a list of 10 symptoms of Parkinsonism (gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, head rotation, glabella tap, tremor, salivation, and akathisia). Severity of each item was rated on a 5-point Likert scale, with a score of 0 (absence of symptoms) to 4 (severe condition). The SAS total score is the sum of the scores of all 10 items, ranging from 0 to 40 where a higher score indicates a severe condition. Population: Safety Sample included all enrolled participants who received at least one dose of IMP. 'Number analyzed' indicates the number of participants with data available for measure analysis.
  score on a scale
    number analyzed (Participants) | 48 | 46 | 94
    (all) | 0.4 (1.9) | 0.2 (0.6) | 0.3 (1.4)
Abnormal Involuntary Movement Scale (AIMS) Total Score [Mean (Standard Deviation); unit: score on a scale] — AIMS is a 12-item scale. First 10 items are rated on Likert 5-point scale: 0 (best) to 4 (worst). Score of 0 depending on specific item, means either "no abnormal Involuntary movement (AIM)" or "no incapacitation due to AIM" or "no awareness of AIM". Item score of 4 means either "severe AIM" or "severe incapacitation due to AIM" or "being aware of, & severe distress caused by AIM". Items 11,12 are related to dental status, taking dichotomous response: 0=no & 1=yes. AIMS movement score is sum of ratings for first 7 items: possible total scores of 0-28, higher score indicates a severe condition. Population: Safety Sample included all enrolled participants who received at least one dose of IMP. 'Number analyzed' indicates the number of participants with data available for measure analysis.
  score on a scale
    number analyzed (Participants) | 48 | 46 | 94
    (all) | 0.06 (0.32) | 0.02 (0.15) | 0.04 (0.25)
Barnes Akathisia Rating Scale (BARS) Score [Mean (Standard Deviation); unit: score on a scale] — BARS consists of 4 items related to akathisia: objective observation of akathisia by the investigator, subjective feelings of restlessness by the participant, subjective distress due to akathisia, and global clinical assessment of akathisia. The first 3 items were rated on a 4-point Likert scale, with a score of 0 (absence of symptoms) to 3 (severe condition) & global clinical assessment was rated on a 6-point scale, with a score of 0 (absence of symptoms) to 5 (severe akathisia). Total score is the sum of the scores of all 4 items, ranging from 0 to 14. Lower scores indicate less symptoms. Population: Safety Sample included all enrolled participants who received at least one dose of IMP. 'Number analyzed' indicates the number of participants with data available for measure analysis.
  score on a scale
    number analyzed (Participants) | 48 | 46 | 94
    (all) | 0.04 (0.20) | 0.09 (0.46) | 0.06 (0.35)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs) Graded By Severity, Serious TEAEs and Trial Discontinuation Due to TEAEs
Description: An AE is any untoward medical occurrence in a clinical trial participant administered a medicinal product that does not necessarily have a causal relationship with the treatment. An SAE: AE that results in the appearance of (or worsening of any pre-existing) undesirable signs, symptoms, or medical conditions i.e. fatal, life-threatening, result in persistent or significant disability/incapacity, constitutes a congenital anomaly/birth defect, and requires inpatient hospitalization or prolongation of existing hospitalization. A TEAE is defined as an AE that started after trial drug treatment; or if the event was continuous from baseline and was worsening, serious, trial drug-related, or resulted in death, discontinuation, interruption, or reduction of trial therapy. TEAEs were graded as, Mild: Discomfort noticed, but no disruption to daily activity, Moderate: Discomfort sufficient to reduce or affect normal daily activity, and Severe: Inability to work or perform normal daily activity.
Time Frame: From the first dose of study drug (in current study) up to 21 days after the last dose of study drug (up to approximately 29 weeks)
Population: Safety Sample included all enrolled participants who received at least one dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Brexpiprazole | Prior Placebo
Number analyzed (Participants) | 49 | 46
Participants
  Participants With TEAEs | 23 | 24
  Participants With Mild TEAEs | 15 | 19
  Participants With Moderate TEAEs | 11 | 12
  Participants With Severe TEAEs | 2 | 2
  Participants With Serious TEAEs | 2 | 1
  Participants With Trial Discontinuations due to TEAEs | 2 | 4

2. Primary Outcome: Number of Participants With Potentially Clinically Relevant Abnormalities in Vital Signs
Description: Vital signs measurements included body weight, body temperature, systolic blood pressure (SBP), diastolic blood pressure (DBP), and heart rate. Blood pressure (i.e., SBP, DBP) and heart rate were measured in the supine and standing positions after the participant had been in each position for at least 3 minutes. The participants were categorized based on the clinically relevant vital sign values as per protocol-predefined criteria. The categories with at least one participant with clinically significant value outside the normal range for vital signs are reported.
Time Frame: Baseline (current study) up to Week 26
Population: Safety Sample included all enrolled participants who received at least one dose of IMP. 'Overall number of participants analyzed' indicates the number of participants with data available for this outcome measure. 'Number analyzed' indicates the number of participants with data available for analysis of the specified parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Brexpiprazole | Prior Placebo
Number analyzed (Participants) | 48 | 46
Participants
  SBP Standing (mmHg): High: number analyzed (Participants) | 47 | 46
  SBP Standing (mmHg): High | 4 | 5
  SBP Supine (mmHg): High | 1 | 5
  DBP Standing (mmHg): Low: number analyzed (Participants) | 47 | 46
  DBP Standing (mmHg): Low | 0 | 1
  DBP Standing (mmHg): High: number analyzed (Participants) | 47 | 46
  DBP Standing (mmHg): High | 2 | 1
  DBP Supine (mmHg): Low | 1 | 1
  DBP Supine (mmHg): High | 1 | 3
  Heart Rate Standing (beats/min): High: number analyzed (Participants) | 47 | 46
  Heart Rate Standing (beats/min): High | 10 | 4
  Heart Rate Supine (beats/min): Low | 1 | 0
  Heart Rate Supine (beats/min): High | 3 | 1
  Body Temperature | 0 | 0

3. Primary Outcome: Number of Participants With Potentially Clinically Relevant Electrocardiogram (ECG) Abnormalities
Description: Twelve-lead ECG recordings were obtained after the participant was supine and at rest for at least 5 minutes. Criteria for identifying ECG measurements of potential clinical relevance included Rate: Tachycardia (Vent ≥110 beats per minute [bpm]; increase ≥15bpm), Bradycardia (Vent ≤ 60bpm; decrease ≥15bpm); Rhythm: Sinus tachycardia (≥ 110bpm; an increase of ≥15 bpm), Sinus bradycardia (≤ 60bpm; a decrease of ≥15 bpm), Supraventricular premature beat (not present at baseline and present post-baseline), Conduction: Right bundle branch block (not present at baseline and present post-baseline) and ST/T Morphology: Symmetrical T-Wave Inversion (not present at baseline and present post-baseline). The categories with at least one participant with clinically relevant ECG abnormalities are reported.
Time Frame: Baseline (current study) up to Week 26
Population: Safety Sample included all enrolled participants who received at least one dose of IMP. 'Overall number of participants analyzed' indicates the number of participants with data available for this outcome measure. 'Number analyzed' indicates the number of participants with data available for the analysis of the specified parameter.
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Brexpiprazole | Prior Placebo
Number analyzed (Participants) | 45 | 43
Participants
  Rate: Tachycardia: number analyzed (Participants) | 43 | 41
  Rate: Tachycardia | 1 | 2
  Rate: Bradycardia: number analyzed (Participants) | 43 | 41
  Rate: Bradycardia | 1 | 0
  Rhythm: Sinus Tachycardia: number analyzed (Participants) | 43 | 41
  Rhythm: Sinus Tachycardia | 1 | 2
  Rhythm: Sinus Bradycardia: number analyzed (Participants) | 43 | 41
  Rhythm: Sinus Bradycardia | 1 | 0
  Rhythm: Supraventricular Premature Beat: number analyzed (Participants) | 44 | 43
  Rhythm: Supraventricular Premature Beat | 1 | 0
  Conduction: Right Bundle Branch Block | 0 | 1
  ST/T Morphology: Symmetrical T-Wave Inversion | 0 | 1

4. Primary Outcome: Number of Participants With Potentially Clinically Relevant Laboratory Test Abnormalities
Description: Laboratory assessments included - serum chemistry including prolactin and thyrotropin, hematology, and urinalysis. Number of participants with potentially clinically relevant laboratory test abnormalities were reported as per criteria defined in SAP. The categories with at least one participant with clinically relevant value outside the normal range for laboratory assessments are reported.
Time Frame: Baseline (current study) up to Week 26
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Brexpiprazole | Prior Placebo
Number analyzed (Participants) | 42 | 42
Participants
  Activated Partial Thromboplastin Time (sec): High: number analyzed (Participants) | 39 | 34
  Activated Partial Thromboplastin Time (sec): High | 6 | 2
  Alanine Aminotransferase (U/L): High: number analyzed (Participants) | 41 | 42
  Alanine Aminotransferase (U/L): High | 0 | 2
  Aspartate Aminotransferase (U/L): High | 0 | 1
  Bicarbonate (mEq/L): Low: number analyzed (Participants) | 41 | 42
  Bicarbonate (mEq/L): Low | 14 | 15
  Bilirubin (mg/dL): Low: number analyzed (Participants) | 36 | 31
  Bilirubin (mg/dL): Low | 10 | 8
  Bilirubin (mg/dL): High: number analyzed (Participants) | 36 | 31
  Bilirubin (mg/dL): High | 0 | 1
  Calcium (mg/dL): Low | 0 | 1
  Chloride (mEq/L): High: number analyzed (Participants) | 42 | 41
  Chloride (mEq/L): High | 2 | 0
  Cortisol (ug/dL): Low: number analyzed (Participants) | 36 | 35
  Cortisol (ug/dL): Low | 7 | 9
  Creatinine (mg/dL): High | 1 | 0
  Glucose (mg/dL): Low | 0 | 1
  Glucose (mg/dL): High | 1 | 0
  Potassium (mEq/L): High: number analyzed (Participants) | 42 | 41
  Potassium (mEq/L): High | 1 | 3
  Sodium (mEq/L): High: number analyzed (Participants) | 42 | 41
  Sodium (mEq/L): High | 2 | 0
  Eosinophils/Leukocytes (%): High: number analyzed (Participants) | 41 | 42
  Eosinophils/Leukocytes (%): High | 2 | 3
  Hematocrit (%): Low: number analyzed (Participants) | 41 | 42
  Hematocrit (%): Low | 0 | 1
  Hematocrit (%): High: number analyzed (Participants) | 41 | 42
  Hematocrit (%): High | 1 | 0
  Hemoglobin (g/dL): Low: number analyzed (Participants) | 41 | 42
  Hemoglobin (g/dL): Low | 1 | 0
  Hemoglobin A1C (%): High: number analyzed (Participants) | 42 | 41
  Hemoglobin A1C (%): High | 2 | 4
  Leukocytes (10^9/L): Low: number analyzed (Participants) | 41 | 42
  Leukocytes (10^9/L): Low | 6 | 2
  Leukocytes (10^9/L): High: number analyzed (Participants) | 41 | 42
  Leukocytes (10^9/L): High | 0 | 1
  Neutrophils (10^9/L): High: number analyzed (Participants) | 41 | 42
  Neutrophils (10^9/L): High | 0 | 2
  Neutrophils/Leukocytes (%): Low: number analyzed (Participants) | 41 | 42
  Neutrophils/Leukocytes (%): Low | 8 | 2
  Neutrophils/Leukocytes (%): High: number analyzed (Participants) | 41 | 42
  Neutrophils/Leukocytes (%): High | 0 | 2
  Platelets (10^9/L): High: number analyzed (Participants) | 41 | 42
  Platelets (10^9/L): High | 1 | 1
  Prothrombin Intl. Normalized Ratio: High: number analyzed (Participants) | 39 | 34
  Prothrombin Intl. Normalized Ratio: High | 5 | 2
  Prothrombin Time (sec): High: number analyzed (Participants) | 39 | 34
  Prothrombin Time (sec): High | 3 | 2
  Protein, Urine: Low: number analyzed (Participants) | 42 | 39
  Protein, Urine: Low | 12 | 11
  Protein, Urine: High: number analyzed (Participants) | 42 | 39
  Protein, Urine: High | 10 | 11
  Prolactin (ng/mL): Low | 3 | 4
  Prolactin (ng/mL): High | 1 | 2
  Thyrotropin (uIU/mL): High | 2 | 0

5. Primary Outcome: Number of Participants With Potentially Clinically Relevant Abnormal Physical Examination Values
Description: Physical examination included measurement of height and the examination of the head, ears, eyes, nose, and throat (HEENT); thorax; abdomen; urogenital; extremities; neurological; and skin and mucosae. Participants with abnormal values, as assessed by the investigator were reported.
Time Frame: Baseline (current study) up to Week 26
Population: Safety Sample included all enrolled participants who received at least one dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Brexpiprazole | Prior Placebo
Number analyzed (Participants) | 49 | 46
Participants | 6 | 4

6. Primary Outcome: Number of Participants With Suicidality as Measured by Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: Suicidality as defined as at least one occurrence of suicidal ideation or suicidal behavior, was assessed using C-SSRS. The assessment included "yes" or "no" responses for 5 questions, each related to suicidal ideation (wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods, active suicidal ideation with some intent, active suicidal ideation with specific plan) & suicidal behavior (preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt, suicide). Numeric ratings were provided for suicidal ideation: Score range of 1 (wish to be dead) to 5 (active suicidal ideation with specific plan and intent), higher total scores indicate more suicidal ideation; Suicidal behavior: Score range of 0 (no suicidal behavior) to 4 (actual suicide attempt), higher total scores indicate more suicidal behavior. Number of participants with at least one occurrence of suicidal ideation or suicidal behavior was reported.
Time Frame: Baseline (current study) up to Week 26
Population: Safety Sample included all enrolled participants who received at least one dose of IMP.
Measure: Count of Participants; unit: Participants
Arm/Group | Prior Brexpiprazole | Prior Placebo
Number analyzed (Participants) | 49 | 46
Participants | 4 | 2

7. Primary Outcome: Change From Baseline in Simpson Angus Scale (SAS) Total Score at Week 2
Description: SAS was used to evaluate extrapyramidal symptoms (EPS). The SAS consists of a list of 10 symptoms of Parkinsonism (gait, arm dropping, shoulder shaking, elbow rigidity, wrist rigidity, head rotation, glabella tap, tremor, salivation, and akathisia). Severity of each item was rated on a 5-point Likert scale, with a score of 0 (absence of symptoms) to 4 (severe condition). The SAS total score is the sum of the scores of all 10 items, ranging from 0 to 40 where a higher score indicates a severe condition. Negative change from baseline indicates absence of symptoms.
Time Frame: Baseline and Week 2
Population: Safety Sample included all enrolled participants who received at least one dose of IMP. 'Overall number of participants analyzed' indicates the number of participants with data available for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior Brexpiprazole | Prior Placebo
Number analyzed (Participants) | 45 | 41
score on a scale | -0.0 (0.5) | 0.0 (0.5)

8. Primary Outcome: Change From Baseline in SAS Total Score at Week 14
Description: as for outcome 7
Time Frame: Baseline and Week 14
Population: Safety Sample included all enrolled participants who received at least one dose of IMP. 'Overall Number of Participants Analyzed' indicates the number of participants with data available for outcome measure analysis at specified time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior Brexpiprazole | Prior Placebo
Number analyzed (Participants) | 38 | 37
score on a scale | -0.1 (0.7) | 0.2 (0.6)

9. Primary Outcome: Change From Baseline in SAS Total Score at Week 26
Description: as for outcome 7
Time Frame: Baseline and Week 26
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior Brexpiprazole | Prior Placebo
Number analyzed (Participants) | 36 | 28
score on a scale | -0.1 (0.9) | -0.0 (0.2)

10. Primary Outcome: Change From Baseline in Abnormal Involuntary Movement Scale (AIMS) Total Score at Week 2
Description: The AIMS is a 12-item scale. The first 10 items are rated on a Likert 5-point scale from 0 to 4 (0 = best, 4 = worst). An item score of 0, depending on specific item, means either "no abnormal Involuntary movement (AIM)" or "no incapacitation due to AIM" or "no awareness of AIM". An item score of 4 means either "severe AIM" or "severe incapacitation due to AIM" or "being aware of, and severe distress caused by AIM". Items 11 and 12 are related to dental status, taking dichotomous response: 0 = no and 1 = yes. AIMS movement score is the sum of the ratings for the first seven items with possible total scores of 0 to 28, where a higher score indicates a severe condition.
Time Frame: Baseline and Week 2
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior Brexpiprazole | Prior Placebo
Number analyzed (Participants) | 45 | 43
score on a scale | 0.0 (0.00) | 0.14 (1.08)

11. Primary Outcome: Change From Baseline in AIMS Total Score at Week 14
Description: as for outcome 10
Time Frame: Baseline and Week 14
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior Brexpiprazole | Prior Placebo
Number analyzed (Participants) | 40 | 38
score on a scale | 0.0 (0.00) | 0.16 (1.15)

12. Primary Outcome: Change From Baseline in AIMS Total Score at Week 26
Description: The AIMS is a 12-item scale. The first 10 items are rated on a Likert 5-point scale from 0 to 4 (0 = best, 4 = worst). An item score of 0, depending on specific item, means either "no abnormal Involuntary movement (AIM)" or "no incapacitation due to AIM" or "no awareness of AIM". An item score of 4 means either "severe AIM" or "severe incapacitation due to AIM" or "being aware of, and severe distress caused by AIM". Items 11 and 12 are related to dental status, taking dichotomous response: 0 = no and 1 = yes. AIMS movement score is the sum of the ratings for the first seven items with possible total scores of 0 to 28, where a higher score indicates a severe condition. A negative change from baseline indicates less symptoms.
Time Frame: Baseline and Week 26
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior Brexpiprazole | Prior Placebo
Number analyzed (Participants) | 36 | 28
score on a scale | 0.00 (0.00) | -0.04 (0.19)

13. Primary Outcome: Change From Baseline in Barnes Akathisia Rating Scale (BARS) Score at Week 2
Description: The BARS consists of 4 items related to akathisia: objective observation of akathisia by the investigator, subjective feelings of restlessness by the participant, subjective distress due to akathisia, and global clinical assessment of akathisia. The first 3 items were rated on a 4-point Likert scale, with a score of 0 (absence of symptoms) to 3 (severe condition) and the global clinical assessment was rated on a 6-point scale, with a score of 0 (absence of symptoms) to 5 (severe akathisia). Total score is the sum of the scores of all 4 items, ranging from 0 to 14. Lower scores indicate less symptoms.
Time Frame: Baseline and Week 2
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior Brexpiprazole | Prior Placebo
Number analyzed (Participants) | 45 | 43
score on a scale | 0.02 (0.26) | 0.05 (0.30)

14. Primary Outcome: Change From Baseline in BARS Score at Week 14
Description: The BARS consists of 4 items related to akathisia: objective observation of akathisia by the investigator, subjective feelings of restlessness by the participant, subjective distress due to akathisia, and global clinical assessment of akathisia. The first 3 items were rated on a 4-point Likert scale, with a score of 0 (absence of symptoms) to 3 (severe condition) and the global clinical assessment was rated on a 6-point scale, with a score of 0 (absence of symptoms) to 5 (severe akathisia). Total score is the sum of the scores of all 4 items, ranging from 0 to 14. Lower scores indicate less symptoms and negative change from baseline indicate less symptoms.
Time Frame: Baseline and Week 14
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior Brexpiprazole | Prior Placebo
Number analyzed (Participants) | 40 | 38
score on a scale | -0.05 (0.22) | 0.05 (0.40)

15. Primary Outcome: Change From Baseline in BARS Score at Week 26
Description: as for outcome 14
Time Frame: Baseline and Week 26
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior Brexpiprazole | Prior Placebo
Number analyzed (Participants) | 36 | 28
score on a scale | 0.00 (0.24) | -0.04 (0.19)

16. Primary Outcome: Percentage of Participants With Potentially Clinically Relevant Changes in Weight up to Week 14
Description: Percentage of participants who had significant weight gain (≥ 7% increase in body weight relative to baseline) and significant weight loss (≥ 7% decrease in body weight relative to baseline) were reported.
Time Frame: Baseline up to Week 14
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Prior Brexpiprazole | Prior Placebo
Number analyzed (Participants) | 40 | 37
percentage of participants
  Weight Gain >= 7% | 45.0 | 48.6
  Weight Loss >= 7% | 0.0 | 0.0

17. Primary Outcome: Percentage of Participants With Potentially Clinically Relevant Changes in Weight up to Week 26
Description: as for outcome 16
Time Frame: Baseline up to Week 26
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Prior Brexpiprazole | Prior Placebo
Number analyzed (Participants) | 39 | 30
percentage of participants
  Weight Gain >= 7% | 71.8 | 76.7
  Weight Loss >= 7% | 0.0 | 3.3

18. Primary Outcome: Time to Discontinuation Due to AE
Description: The time to discontinuation due to AE was defined as the total number of days between the enrolment date and the discontinuation date. The time to discontinuation was analyzed using the Kaplan Meier curve.
Time Frame: Baseline (in current study) up to 21 days post last dose of study drug (up to approximately 29 weeks)
Population: as for outcome 7
Measure: Median (Full Range); unit: days
Arm/Group | Prior Brexpiprazole | Prior Placebo
Number analyzed (Participants) | 2 | 4
days | 83 [14 to 152] | 113 [54 to 140]

19. Secondary Outcome: Mean Change From Baseline to Week 26 in Aberrant Behavior Checklist - Irritability (ABC-I) Subscale Score
Description: The ABC is parent-reported rating scale designed to assess treatment effects on problem behavior in participants with intellectual disabilities. The ABC scale has 58 items, which divide into 5 subscales as follows:(1) Irritability, Agitation; (2) Lethargy, Social Withdrawal; (3) Stereotypic Behavior; (4) Hyperactivity, Noncompliance; and (5) Inappropriate Speech. Each of the 58 ABC items is rated on a 4-point scale (0 = not at all a problem; 1=the behavior is a problem, but slight in degree; 2=problem is moderately serious; 3=problem is severe in degree). The Irritability subscale (ABC-I) measures emotional and behavioral symptoms of ASD, including aggression toward others, deliberate self-injuriousness, temper tantrums, & quickly changing moods. ABC-I total score is the sum of the ratings over 15 ABC items. Individual scores were summed, thus the ABC-I total score ranges from 0 to 45. Higher scores represent the worst condition. Negative change from baseline indicates less symptoms.
Time Frame: Baseline (current study), Week 26
Population: Efficacy Sample included all participants in the Safety Sample who had a baseline assessment and at least one post-baseline assessment of the ABC-I subscale score. 'Overall number of participants analyzed' indicates the number of participants with data available for this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior Brexpiprazole | Prior Placebo
Number analyzed (Participants) | 35 | 27
score on a scale | -5.47 (8.06) | -7.00 (8.36)

20. Secondary Outcome: Mean Change From Baseline to Week 26 in Clinical Global Impression - Severity (CGI-S) Scale Score
Description: The CGI-S scale is a clinician-rated assessment that evaluates the severity of a participant's condition with a focus on symptoms of irritability on a 7-point scale. The investigator (or rater) answered the following question: "Considering your total clinical experience with this particular population, how ill was the participant at this time with regard to symptoms of irritability?" Response choices were 0 = not assessed; 1 = normal, not at all ill; 2 = borderline ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; and 7 = among the most extremely ill patients. The total score ranges from 0 to 7, where higher scores indicate worse condition. A negative change from baseline indicates less symptoms.
Time Frame: Baseline (current study), Week 26
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prior Brexpiprazole | Prior Placebo
Number analyzed (Participants) | 36 | 28
score on a scale | -0.78 (0.99) | -0.68 (0.94)

ADVERSE EVENTS:
Time Frame: From the first dose of study drug (in current study) up to 21 days after the last dose of study drug (up to approximately 29 weeks)
Description: Safety Sample included all enrolled participants who received at least one dose of IMP.
Arm/Group | Prior Brexpiprazole | Prior Placebo
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/46
Serious Adverse Events (participants affected / at risk) | 2/49 | 1/46
Other Adverse Events (participants affected / at risk) | 17/49 | 11/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prior Brexpiprazole (N=49) | Prior Placebo (N=46)
Dyskinesia (Nervous system disorders) | 1 | 0
Affective Disorder (Psychiatric disorders) | 0 | 1
Suicidal Ideation (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prior Brexpiprazole (N=49) | Prior Placebo (N=46)
Gastroenteritis (Infections and infestations) | 3 | 0
Viral Influenza (Infections and infestations) | 4 | 0
Weight Increased (Investigations) | 5 | 8
Increased Appetite (Metabolism and nutrition disorders) | 2 | 4
Somnolence (Nervous system disorders) | 5 | 1
Irritability (Psychiatric disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/39/NCT04258839/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-08): https://cdn.clinicaltrials.gov/large-docs/39/NCT04258839/SAP_001.pdf